CLINICAL TRIAL: NCT02300727
Title: A Phase I/II Study to Determine the Safety and Efficacy of Curcumin in Patients With Oral Mucositis Secondary to Chemotherapy
Brief Title: Study to See How Safe Curcumin is and How Well it Works When Used to Treat Mucositis in Patients Getting Chemotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Protocol failed to accrue sufficient subject to complete meaningful analysis.
Sponsor: Amy Beres (Other)
Responsible Party: Sponsor-Investigator, Amy Beres, Oncology Physician, Aurora BayCare Medical Center
Organization: Aurora BayCare Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Curcumin:I/II
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Mucositis
Keywords: Mucositis; Neoplasms; CANCER; Curcumin; Drug Therapy; ANTINEOPLASTIC AGENTS
MeSH Terms: conditions — Mucositis; Neoplasms | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mouthwash-standard pharmacy preparation (Active Comparator): Standard mouth wash preparation administered by ingested mouth rinse three times per day.
  The standard mouth rinse contains 40% Benadryl, 40% Maalox, and 20% of 1% Viscous Lidocaine.
  Interventions: Drug: Mouthwash-standard pharmacy preparation
- Curcumin (Experimental): Curcumin (BCM-95) administered by ingested mouth rinse three times per day. Subjects will be in this arm at the previously determine maximum tolerated dose (MTD).
  Interventions: Drug: Curcumin
- Curcumin-MTD (Other): Curcumin (BCM-95) administered by ingested mouth rinse. A total of 12-15 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participant at each of 4 does levels (0.33g, 1g, 2g, 3g) per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Interventions: Drug: Curcumin-MTD

INTERVENTIONS:
Drug: Curcumin-MTD — 0.33g-3g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
  Other Names: Curcumin; BCM-95; Tumeric
  Arms: Curcumin-MTD
Drug: Mouthwash-standard pharmacy preparation — Standard mouth wash preparation administered by ingested mouth rinse three times per day.
  The standard mouth rinse contains 40% Benadryl, 40% Maalox, and 20% of 1% Viscous Lidocaine.
  Other Names: no other name
  Arms: Mouthwash-standard pharmacy preparation
Drug: Curcumin — After maximum tolerated dose (MTD) is determined, MTD by ingested mouth wash three times per day for 4-6 weeks until mucositis is resolved, disease progression, or unacceptable toxicity develops.
  Other Names: BCM-95; Tumeric
  Arms: Curcumin

SUMMARY:
Oral mucositis is a common side effect from cancer treatment. Patients receiving chemotherapy and radiotherapy can get very painful sores in their mouth that compromise nutrition and oral hygiene as well as increase risk for infection, and can last for weeks. Currently, the only treatment for mucositis is oral hygiene to try to support recovery.

Curcumin (also known as Turmeric) is a frequently-used spice in India and Southeast Asia. Studies in cells and animals have shown that it can reduce the amount of bacteria and can prevent inflammation.

In this study, the investigators want to learn if a mouthwash made with curcumin is safe for people to use and if it can help their mucositis.

DETAILED DESCRIPTION:
This is a phase I/II study involving 2 parts; a dose escalation to determine the maximum tolerated dose (MTD) of curcumin and an expansion at the MTD.

Oral mucositis is a common and often debilitating complication associated with cancer treatment. Treatment of mucositis is mainly supportive - oral hygiene is the means of treatment. Curcumin (Turmeric), a frequently-used spice in India and Southeast Asia, can reduce bacterial load and prevent inflammation in cultured epithelial cells and prevent chemotherapy- and radiotherapy-induced mucositis in animal models.

The primary objective of this Phase I/II study is to determine the maximum tolerated dose (MTD) of oral curcumin in patients who have chemotherapy-induced mucositis. The secondary objectives of this study are to determine whether or not oral curcumin has an acceptable safety profile or impacts oral mucositis health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ grade 2 oral mucositis related to chemotherapy for cancer
* Ability to understand and the willingness to review and sign a written informed consent document.
* ≥ 18 years of age
* Willingness to use adequate contraception prior to study entry, for the duration of study participation and for 30 days after the last dose for women of child-bearing potential and men

Exclusion Criteria:

* Current use of therapeutic doses of anticoagulants such as warfarin or antiplatelet agents (prophylactic doses and agents are acceptable)
* Biliary tract obstruction or cholelithiasis
* History of gastric or duodenal ulcers or hyperacidity syndromes
* AST or ALT > 2 x ULN
* Total bilirubin ≥ 2 x ULN
* INR > 1.5
* Previous stem cell transplant (allogeneic or autologous)
* Preexisting oral disease, such as active oral infection, trauma to the oral mucosa or oral - ulceration prior to chemotherapy
* Known allergy/hypersensitivity to curcumin, yellow food coloring, or other members of the - Zingiberaceae (ginger) family
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-02; Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhimant Patel, MD, Principal Investigator — Aurora BayCare Medical Center
Locations (1):
- Aurora BayCare Medical Center, Green Bay, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mouthwash-standard Pharmacy Preparation: Standard mouth wash preparation administered by ingested mouth rinse three times per day.
  The standard mouth rinse contains 40% Benadryl, 40% Maalox, and 20% of 1% Viscous Lidocaine.
  Mouthwash-standard pharmacy preparation: Standard mouth wash preparation administered by ingested mouth rinse three times per day.
  The standard mouth rinse contains 40% Benadryl, 40% Maalox, and 20% of 1% Viscous Lidocaine.
- Curcumin-MTD 0.33g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participant at a dose level of 0.33g per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 0.33g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
- Curcumin-MTD 1g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participant at a dose level of 1g per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 1g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
- Curcumin- MTD 2g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participant at a dose level of 2g per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 2g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
- Curcumin- MTD 3g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participant at a dose level of 3g per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 3g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
Period: Overall Study
Arm/Group | Mouthwash-standard Pharmacy Preparation | Curcumin | Curcumin-MTD 0.33g Dose | Curcumin-MTD 1g Dose | Curcumin- MTD 2g Dose | Curcumin- MTD 3g Dose
Started | 0 | 0 | 3 | 3 | 0 | 0
Completed | 0 | 0 | 3 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Insufficient accrual to this protocol for meaningful analysis.
Groups:
- Curcumin-MTD 0.33g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participant at a dose of 0.33g curcumin per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 0.33g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
- Curcumin-MTD 1g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participant at a dose of 1g curcumin per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 1g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
- Curcumin-MTD 2g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participant at a dose of 2g curcumin per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 2g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
- Curcumin-MTD 3g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participant at a dose of 3g curcumin per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 3g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
- Total: Total of all reporting groups
Arm/Group | Mouthwash-standard Pharmacy Preparation | Curcumin | Curcumin-MTD 0.33g Dose | Curcumin-MTD 1g Dose | Curcumin-MTD 2g Dose | Curcumin-MTD 3g Dose | Total
Number analyzed (Participants) | 0 | 0 | 3 | 3 | 0 | 0 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  |  | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years |  |  | 3 | 3 | 0 | 0 | 6
  >=65 years |  |  | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 2 | 2 | 0 | 0 | 4
  Male |  |  | 1 | 1 | 0 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Number of Participants with Serious and Non-Serious Adverse Events.
Time Frame: reviewed weekly for 4 to 6 weeks
Population: Protocol ended early after failing to enroll sufficiently. Only 6 subjects enrolled, 5 completed, 1 withdrew. Insufficient data to analyze.
Measure: Count of Participants; unit: Participants
Groups:
- Curcumin-MTD 0.33g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participants at a dose of 0.33g curcumin per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 0.33g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
- Curcumin-MTD 1g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participants at a dose of 1g curcumin per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 1g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
- Curcumin- MTD 2g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participants at a dose of 2g curcumin per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 2g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
- Curcumin- MTD 3g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participants at a dose of 3g curcumin per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 3g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
Arm/Group | Mouthwash-standard Pharmacy Preparation | Curcumin | Curcumin-MTD 0.33g Dose | Curcumin-MTD 1g Dose | Curcumin- MTD 2g Dose | Curcumin- MTD 3g Dose
Number analyzed (Participants) | 0 | 0 | 3 | 3 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Change in Toxicities Graded by Health Care Providers Using the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: NA - Protocol ended early after failing to enroll sufficiently. Only 6 subjects enrolled, 5 completed, 1 withdrew. Zero participants analyzed.
Time Frame: Baseline, weekly for 5 to 7 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Change in Subjective Patient Self-assessment of Pain.
Description: NA - Protocol ended early after failing to enroll sufficiently. Only 6 subjects enrolled, 5 completed, 1 withdrew. Insufficient data to analyze
Time Frame: Baseline, weekly for 5 to 7 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change in Subjective Patient Self- Assessment of Oral Mucositis Measured by the Common Terminology Criteria for Adverse Events (CTCAE) and World Health Organization's (WHO's) Oral Toxicity Scale (OTS)
Description: as for outcome 3
Time Frame: Baseline, weekly for 5 to 7 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change in Health Providers Assessment of Oral Mucositis and Healing Time Measured by the Common Terminology Criteria for Adverse Events (CTCAE) and World Health Organization's (WHO's) Oral Toxicity Scale (OTS)
Description: as for outcome 3
Time Frame: Baseline, then weekly for 4 to 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months
Description: Zero enrollments in Curcumin-MTD 2g dose, Curcumin-MTD 3g dose, Mouthwash Standard, and Curcumin groups.
Groups:
- Curcumin-MTD 2g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participants at a dose of 2g curcumin per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 2g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
- Curcumin-MTD 3g Dose: Curcumin (BCM-95) administered by ingested mouth rinse. A total of 3-6 subjects will be in this arm to determine maximum tolerated dose (MTD).
  There will be 3 participants at a dose of 3g curcumin per rinse, three times daily for 4-6 weeks. (additional 3 subjects if a dose-limiting toxicity occurs)
  Curcumin-MTD: 3g by ingested mouth wash three times per day for 4-6 weeks until unacceptable toxicity develops- to determine the maximum tolerated does (MTD).
Arm/Group | Mouthwash-standard Pharmacy Preparation | Curcumin | Curcumin-MTD 0.33g Dose | Curcumin-MTD 1g Dose | Curcumin-MTD 2g Dose | Curcumin-MTD 3g Dose
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/3 | 0/3 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/3 | 0/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/3 | 0/3 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT02300727/Prot_SAP_000.pdf